CLINICAL TRIAL: NCT01068002
Title: Hypertension During Pregnancy: Cardiovascular & Echocardiographic Assessment: CREATION - P (01)
Brief Title: Cardiovascular an Echocardiographic Assessment in Hypertension During Pregnancy
Acronym: CREATION-P
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr. Limor Ilan- Bushari, Ha'Emek Medical Center
Other Study IDs: 071-09-EMC
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy
Keywords: Hypertension Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control, normotensive, pregnancy: Control, normotensive, pregnancy
- hypertension, pregnancy, no treatment: hypertension, pregnancy, no treatment
- hypertension, pregnancy, drug treatment: hypertension, pregnancy, drug treatment

SUMMARY:
Cardiovascular & echocardiographic assessment in pregnant women with hypertension during their pregnancy in comparison to Pregnant normotensive women.

DETAILED DESCRIPTION:
Cardiovascular & echocardiographic assessment in pregnant women with hypertension during their pregnancy in comparison to Pregnant normotensive women. Also,comparing echocardiographic parameters in hypertensive pregnant women being treated with either alfa methyl dopa or labetolol.

ELIGIBILITY:
Inclusion Criteria:

* hypertension during pregnancy: Chronic or pregnancy induced

Exclusion Criteria:

* Inability to sign informed consent

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant Women
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Hypertension impact on cardiovascular echocardiographic parameters and obstetric parameters in pregnant women with or without treatment | 1 year

SECONDARY OUTCOMES:
Primary outcome, Impact of alfa methyl dopa and labetolol on cardiovascular parameters in pregnant women | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Limor I Bushari, Principal Investigator — Heart Institute, Ha'Emek Medical Center
Locations (1):
- Ha'Emek Medical Center, Afula, Israel